CLINICAL TRIAL: NCT00957047
Title: Efficacy and Safety of BIA 2-093 as Adjunctive Therapy for Refractory Partial Seizures in a Double-blind, Randomised, Placebo-controlled, Parallel-group, Multicentre Clinical Trial
Brief Title: Efficacy and Safety Study of BIA 2-093 in Combination With Other Anti-Epileptic Drugs to Treat Partial Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-2093-302
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Results first posted 2013-08-05 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Partial Epilepsy
Keywords: refractory; partial; epilepsy
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — eslicarbazepine acetate; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- ESL 400 mg once daily (Experimental): Eslicarbazepine acetate (ESL) was supplied in 400 mg tablets for Part I
  Interventions: Drug: eslicarbazepine acetate
- ESL 800 mg once daily (Experimental): Eslicarbazepine acetate (ESL) was supplied in 800-mg tablets for Part I
  Interventions: Drug: eslicarbazepine acetate
- ESL 1200 mg once daily (Experimental): Eslicarbazepine acetate (ESL) was supplied in 400-mg and 800-mg tablets for Part I
  Interventions: Drug: eslicarbazepine acetate
- placebo (Placebo Comparator): Placebo tablets matching the 400-mg and 800-mg active substance tablets were supplied
  Interventions: Drug: placebo
- ESL - Part II (Experimental): All patients in Part II (Open-label Extension ) received ESL on an open-label basis, starting at 800 mg once daily.
  Interventions: Drug: ESL - Part II

INTERVENTIONS:
Drug: eslicarbazepine acetate — oral tablets
  Other Names: Zebinix
  Arms: ESL 1200 mg once daily; ESL 400 mg once daily; ESL 800 mg once daily
Drug: placebo — once daily placebo comparator
  Other Names: Sugar pill
  Arms: placebo
Drug: ESL - Part II — Eslicarbazepine acetate was supplied as scored 800-mg tablets for daily oral administration.
  Other Names: Eslicarbazepine acetate (ESL), BIA 2-093
  Arms: ESL - Part II

SUMMARY:
The primary objective of the study is to evaluate the efficacy of eslicarbazepine acetate once-daily at doses of 400 mg, 800 mg and 1200 mg compared with placebo as adjunctive therapy in patients with refractory partial epilepsy over a 12-week maintenance period. Patients who complete Part I may enter a 1-year open-label extension.

DETAILED DESCRIPTION:
Part I was a 22-week parallel-group, randomized, placebo-controlled period (8 weeks baseline, 2 weeks double-blind titration, and 12 weeks maintenance). After completing the baseline period, patients were randomized in a 1:1:1:1 ratio to 1 of the 3 ESL dose levels or to placebo.

Part II was a 1-year open-label extension for patients who had completed Part I. The starting dose was 800 mg once daily and could be titrated up or down at 400-mg intervals between 400 and 1200 mg.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent signed by patient
* aged 18 years or more
* documented diagnosis of simple or complex partial seizures with or without secondary generalisation since at least 12 months prior to screening
* at least 4 partial seizures in each 4 week period during the last 8 weeks prior to screening, currently treated with 1 or 2 AEDs (any except oxcarbazepine and felbamate), in a stable dose regimen during at least 2 months prior to screening (patients using vigabatrin should have been on this medication for at least 1 year with no deficit in visual field identified)
* excepting epilepsy, patient is judged to be in general good health based on medical history, physical examination and laboratory tests
* post-menopausal or otherwise incapable of becoming pregnant by reason of surgery or tubal ligation; in case of woman of childbearing potential, patient must present a serum beta-hCG test consistent with a non-gravid state and agree to remain abstinent or use reliable contraception (oral contraception should be combined with a barrier method

Exclusion Criteria:

* only simple partial seizures with no motor symptomatology (classified as A2-4 according to the International Classification of Epileptic Seizures) that are not video-EEG documented
* primarily generalised epilepsy
* known rapid progressive neurological disorder; history of status epilepticus or cluster seizures (i.e., 3 or more seizures within 30 minutes) within the 3 months prior to screening
* seizures of psychogenic origin within the last 2 years
* history of schizophrenia or suicide attempt
* currently on or with exposure to felbamate or oxcarbazepine more within one month of screening
* using benzodiazepines on more than on an occasional basis (except when used chronically as AED)
* previous use of ESL or participation in a clinical study with ESL
* known hypersensitivity to carbamazepine, oxcarbazepine or chemically related substances
* history of abuse of alcohol, drugs or medications within the last 2 years
* uncontrolled cardiac, renal, hepatic, endocrine, gastrointestinal, metabolic, haematological or oncology disorder
* second or third-degree atrioventricular blockade not corrected with a pacemaker
* relevant clinical laboratory abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2004-07; Primary Completion 2006-08 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elinor Ben-Menachem, MD, Principal Investigator — Sahlgren University Hospital, Göteborg, Sweden; Alberto Alain Gabbai, MD, Principal Investigator — Rua Pedro de Toledo 655, Vila Clemento, Sao Paulo, Brazil
Locations (1):
- Bial - Portela & Cª, S.A., Trofa, Coronado (S.Romão E S. Mamede), Portugal

REFERENCES:
- [Derived] Andermann E, Rosenfeld W, Penovich P, Rogin J, Cendes F, Carreno M, Ramsay RE, Ben-Menachem E, Gama H, Rocha F, Soares-da-Silva P, Tosiello R, Blum D, Grinnell T. Comparative analysis of the safety and tolerability of eslicarbazepine acetate in older (>/=60 years) and younger (18-59 years) adults. Epilepsy Res. 2021 Jan;169:106478. doi: 10.1016/j.eplepsyres.2020.106478. Epub 2020 Oct 10. PMID 33338829

RESULTS

PARTICIPANT FLOW:
Recruitment Details: STUDY DATES:
  PART I - From: 01 Sep 2004 To: 19 Dec 2006; PART II - From: 02 February 2005 To: 29 January 2008 Patients were screened at 46 sites in 13 countries for Part I and Patients from 42 sites in 12 countries continued in part II.;
Pre-assignment Details: Part I was a 22-week parallel-group, randomized, placebo controlled period. After completing the baseline period, patients were randomized in a 1:1:1:1 ratio to 1 of the 3 ESL dose levels or to placebo. For Part I 400 patients were planned; of 503 patients screened, 395 were randomized. 325 patients who completed Part I were enrolled in Part II.
Groups:
- Placebo: placebo : once daily placebo comparator
- ESL 400 mg Once Daily; ESL 800 mg Once Daily; ESL 1200 mg Once Daily: eslicarbazepine acetate : oral tablets
- ESL - Part II: All patients in Part II received ESL on an open-label basis, starting at 800 mg once daily.
Period: PART I
Arm/Group | Placebo | ESL 400 mg Once Daily | ESL 800 mg Once Daily | ESL 1200 mg Once Daily | ESL - Part II
Started | 100 | 96 | 101 | 98 | 0
Randomized/Safety Population | 100 | 96 | 101 | 98 | 0
Intention-to-treat (ITT) Population | 100 | 96 | 100 | 97 | 0
Per-Protocol Population | 81 | 70 | 75 | 54 | 0
Completed | 94 | 83 | 80 | 68 | 0
Not Completed | 6 | 13 | 21 | 30 | 0
Period: PART II
Arm/Group | Placebo | ESL 400 mg Once Daily | ESL 800 mg Once Daily | ESL 1200 mg Once Daily | ESL - Part II
Started | 0 | 0 | 0 | 0 | 325 (325 patients who completed Part I were enrolled in Part II.)
Terminated Prematurely | 0 | 0 | 0 | 0 | 102 (Terminated Prematurely during 1-year Open-Label Period)
Completed | 0 | 0 | 0 | 0 | 223
Not Completed | 0 | 0 | 0 | 0 | 102

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ESL 1200 mg Once Daily | ESL 400 mg Once Daily | ESL 800 mg Once Daily | Placebo | Total
Number analyzed (Participants) | 98 | 96 | 101 | 100 | 395
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 98 | 96 | 101 | 98 | 393
  >=65 years | 0 | 0 | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 57 | 50 | 48 | 201
  Male | 52 | 39 | 51 | 52 | 194

OUTCOME MEASURES:

1. Primary Outcome: PART I - Seizure Frequency
Description: The primary efficacy endpoint is the natural log transformation of the seizure frequency per 4 weeks. The primary efficacy analysis was based on the ITT population. Efficacy analyses were performed chiefly using data from the 12-week maintenance period in Part I of the study. The primary efficacy variable is the ln transformation of the seizure frequency per 4 weeks. Seizure frequency was compared between each active treatment group and the placebo group using an ANCOVA that models seizure frequency as a function of baseline seizure frequency and treatment.
Time Frame: 12-week maintenance period
Population: The primary efficacy analysis was an ANCOVA that assessed reduction in seizure frequency per 4 weeks for the ITT population during the 12-week maintenance period
Measure: Least Squares Mean (95% Confidence Interval); unit: ln (Seizures) per 4 weeks
Arm/Group | ESL 1200 mg Once Daily | ESL 400 mg Once Daily | ESL 800 mg Once Daily | Placebo
Number analyzed (Participants) | 97 | 96 | 100 | 100
ln (Seizures) per 4 weeks | 7 [6.0 to 8.1] | 8.7 [7.7 to 9.9] | 7.1 [6.2 to 8.2] | 9.8 [8.7 to 11.1]

2. Primary Outcome: PART II - Nº of Treatment-Emergent Adverse Events (TEAE)
Description: Safety assessments were based primarily on AEs (Number of patients who experienced at least one AEs), and on whether these were related to the study medication, were serious, led to permanent discontinuation of study participation, or led to death.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | TEAE | TEAE With Onset Within the 1st 4 Weeks | TEAE With Onset After 1st 4 Weeks | Treatment-related TEAE | TEAE Leading to Discontinuation | Serious TEAE | TEAE Leading to Death
Number analyzed (Participants) | 325 | 325 | 325 | 325 | 325 | 325 | 325
participants | 270 | 151 | 240 | 194 | 37 | 28 | 3

ADVERSE EVENTS:
Groups:
- Placebo; ESL 400 mg; ESL 800 mg; ESL 1200 mg: Tablets; oral route
- ESL PART II: All patients in Part II received ESL
Arm/Group | Placebo | ESL 400 mg | ESL 800 mg | ESL 1200 mg | ESL PART II
Serious Adverse Events (participants affected / at risk) | 0/100 | 4/96 | 6/101 | 2/98 | 28/325
Other Adverse Events (participants affected / at risk) | 59/100 | 75/96 | 84/101 | 78/98 | 270/325
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=100) | ESL 400 mg (N=96) | ESL 800 mg (N=101) | ESL 1200 mg (N=98) | ESL PART II (N=325)
Acute psychosis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Appendix disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1
Asthenia (General disorders) | 0 | 0/0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 3
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Diplopia (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0
Drowning (General disorders) | 0 | 0 | 0 | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1
Dyskinesia oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0
Follicle centre lymphoma, follicular grade I, II, III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1
Grand mal convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hepatic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0
Insulinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0/0 | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Monocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Ovarian mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0
Schizoaffective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 1
Vasculitis cerebral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=100) | ESL 400 mg (N=96) | ESL 800 mg (N=101) | ESL 1200 mg (N=98) | ESL PART II (N=325)
Coordination abnormal (Nervous system disorders) | 5 (5) | 5 (5) | 13 (13) | 11 (11) | 28
Diplopia (Eye disorders) | 4 (4) | 8 (8) | 15 (15) | 10 (10) | 28
Dizziness (Nervous system disorders) | 10 (10) | 22 (22) | 30 (30) | 43 (43) | 86
Fatigue (General disorders) | 5 (5) | 4 (4) | 5 (5) | 7 (7) | 0
Headache (Nervous system disorders) | 9 (9) | 12 (12) | 15 (15) | 19 (19) | 51
Nausea (Gastrointestinal disorders) | 4 (4) | 8 (8) | 12 (12) | 15 (15) | 21
Somnolence (Nervous system disorders) | 17 (17) | 15 (15) | 17 (17) | 21 (21) | 39
Vision blurred (Eye disorders) | 2 (2) | 7 (7) | 8 (8) | 7 (7) | 17
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4) | 13 (13) | 10 (10) | 22
Blood pressure diastolic decreased (Investigations) | 0 | 0 | 0 | 0 | 28
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 20
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other